CLINICAL TRIAL: NCT03425396
Title: A Randomized, Double-Blinded, Adaptive Phase 2 Study to Evaluate the Safety and Efficacy of Oral Omadacycline and Oral Nitrofurantoin in the Treatment of Female Adults With Cystitis
Brief Title: Oral Omadacycline vs. Oral Nitrofurantoin for the Treatment of Cystitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTK0796-UUTI-17201
Record Dates: First submitted 2017-12-28; First posted 2018-02-07 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Uncomplicated Urinary Tract Infection; Cystitis
MeSH Terms: conditions — Cystitis | interventions — omadacycline; Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Omadacycline 300/300 once every 24 hours (Experimental): Participants received omadacycline 300 milligrams orally, once every 12 hours, fed on Day 1 and omadacycline 300 milligrams orally, once every 24 hours on Days 2 through 7. Odd doses on Days 2 to 7 were administered in a fasted state. Even doses on Days 2 to 7 were administered approximately 2 hours following a light meal.
  Interventions: Drug: Omadacycline tablets
- Omadacycline 450/300 once every 24 hours (Experimental): Participants received omadacycline 450 milligrams orally, once every 12 hours, fed on Day 1 and omadacycline 300 milligrams orally, once every 24 hours on Days 2 through 7. Odd doses on Days 2 to 7 were administered in a fasted state. Even doses on Days 2 to 7 were administered approximately 2 hours following a light meal.
  Interventions: Drug: Omadacycline tablets
- Omadacycline 450/450 once every 24 hours (Experimental): Participants received omadacycline 450 milligrams orally, once every 12 hours, fed on Day 1 and omadacycline 450 milligrams orally, once every 24 hours on Days 2 through 7. Odd doses on Days 2 to 7 were administered in a fasted state. Even doses on Days 2 to 7 were administered approximately 2 hours following a light meal.
  Interventions: Drug: Omadacycline tablets
- Omadacycline 450/450 once every 12 hours (Experimental): Participants received omadacycline 450 milligrams orally, once every 12 hours, fed on Day 1 and omadacycline 450 milligrams orally, once every 12 hours on Days 2 through 7. Odd doses on Days 2 to 7 were administered in a fasted state. Even doses on Days 2 to 7 were administered approximately 2 hours following a light meal.
  Interventions: Drug: Omadacycline tablets
- Nitrofurantoin 100/100 once every 12 hours (Active Comparator): Participants received nitrofurantoin 100 milligrams orally, once every 12 hours, fed on Day 1 and nitrofurantoin 100 milligrams orally, once every 12 hours on Days 2 through 7. Odd doses on Days 2 to 7 were administered in a fasted state. Even doses on Days 2 to 7 were administered approximately 2 hours following a light meal.
  Interventions: Drug: Nitrofurantoin capsules

INTERVENTIONS:
Drug: Omadacycline tablets — Oral Omadacycline
  Arms: Omadacycline 300/300 once every 24 hours; Omadacycline 450/300 once every 24 hours; Omadacycline 450/450 once every 12 hours; Omadacycline 450/450 once every 24 hours
Drug: Nitrofurantoin capsules — Oral Nitrofurantoin
  Arms: Nitrofurantoin 100/100 once every 12 hours

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of oral omadacycline as compared to oral nitrofurantoin in the treatment of female adults with cystitis.

DETAILED DESCRIPTION:
Participants were randomized to receive 7 days of treatment of either omadacycline or nitrofurantoin. The End of Treatment visit, Post Therapy Evaluation visit, and Final Follow-up visit was planned within 2 days following the last dose of study drug, on Day 14 (+/- 2 days) after the first dose of study drug, and within 30 to 37 days following the first dose of study drug, respectively. The study followed a double-dummy design. To maintain the study blinding, participants assigned to omadacycline received active omadacycline tablets and over-encapsulated nitrofurantoin placebo tablets. Participants assigned to the nitrofurantoin arm received omadacycline placebo tablets and over-encapsulated active nitrofurantoin capsules.

ELIGIBILITY:
Inclusion Criteria:

* Female participants, age 18 or older who have signed the informed consent form
* Must have a qualifying uncomplicated urinary tract infection
* Participants must not be pregnant at the time of enrollment
* Must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

* Males
* Evidence of complicated urinary tract infection (UTI), upper UTI, vaginitis, or sexually transmitted infection
* Evidence of significant immunological disease
* Has received an investigational drug within the past 30 days
* Participants who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 225 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Site 106, Chula Vista, California
  - Site 101, La Mesa, California
  - Site 109, Los Angeles, California
  - Site 114, Aventura, Florida
  - Site 102, DeLand, Florida
  - Site 103, Hialeah, Florida
  - Site 125, Jacksonville, Florida
  - Site 121, Miami, Florida
  - Site 130, Miami, Florida
  - Site 115, Miami, Florida
  - Site 127, Miami Springs, Florida
  - Site 126, Orlando, Florida
  - Site 113, Newton, Kansas
  - Site 110, Wichita, Kansas
  - Site 112, Omaha, Nebraska
  - Site 132, Las Vegas, Nevada
  - Site 108, Las Vegas, Nevada
  - Site 122, Berlin, New Jersey
  - Site 118, Raleigh, North Carolina
  - Site 104, Jackson, Tennessee
  - Site 105, Smyrna, Tennessee
  - Site 131, Houston, Texas
  - Site 120, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Started | 55 | 54 | 54 | 8 | 54
Completed End of Treatment Visit | 53 | 52 | 51 | 7 | 53
Completed Post-therapy Evaluation Visit | 53 | 49 | 51 | 7 | 54
Completed Final Follow-up Visit | 53 | 47 | 51 | 7 | 53
Completed | 53 | 47 | 51 | 7 | 53
Not Completed | 2 | 7 | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 5 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population consisted of all randomized participants regardless of whether or not the participant received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours | Total
Number analyzed (Participants) | 55 | 54 | 54 | 8 | 54 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (17.05) | 47.4 (15.70) | 45.0 (15.49) | 37.5 (13.60) | 45.5 (17.82) | 45.5 (16.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 54 | 8 | 54 | 225
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 47 | 43 | 7 | 47 | 191
  Not Hispanic or Latino | 8 | 7 | 11 | 1 | 7 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1 | 2
  Black or African American | 2 | 1 | 4 | 2 | 4 | 13
  White | 52 | 52 | 48 | 6 | 47 | 205
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the Post Therapy Evaluation (PTE) Visit (ITT Population)
Description: Clinical response was determined by the investigator at the PTE visit by assessing whether or not the participant met the clinical outcome of Clinical Success, Clinical Failure, or Indeterminate. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the PTE visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection or reappearance of signs and symptoms at or before the PTE visit such that use of additional systemic antimicrobial therapy for the current infection was required. The clinical outcome was deemed as Indeterminate when the PTE visit was not completed.
Time Frame: Day 14 (A PTE occurred on Day 14 ± 2 days after the participant's first dose of study drug)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 55 | 54 | 54 | 8 | 54
Participants
  Clinical Success | 48 | 42 | 46 | 7 | 49
  Clinical Failure | 5 | 6 | 5 | 0 | 5
  Indeterminate | 2 | 6 | 3 | 1 | 0
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -3.5, 95% CI 2-sided [-16.8 to 9.6] — Point estimate and exact 95% confidence intervals for difference from nitrofurantoin (omadacycline minus nitrofurantoin) in clinical success rate was estimated
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -13.0, 95% CI 2-sided [-27.4 to 1.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -5.6, 95% CI 2-sided [-19.6 to 7.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -3.2, 95% CI 2-sided [-44.1 to 14.7] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the End of Treatment (EOT) Visit (ITT Population)
Description: Clinical response was determined by the investigator at the EOT visit by assessing whether or not the participant met the clinical outcome of Clinical Success, Clinical Failure. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the EOT visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection at the EOT visit such that use of additional systemic antimicrobial therapy for the current infection was required. The clinical outcome was deemed as Indeterminate when the EOT visit was not completed.
Time Frame: EOT visit (within 1 to 2 days following the last dose of study drug i.e. up to approximately 9 days)
Population: The ITT Population consisted of all randomized participants regardless of whether or not the participant received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 55 | 54 | 54 | 8 | 54
Participants
  Clinical Success | 49 | 47 | 49 | 7 | 49
  Clinical Failure | 4 | 5 | 2 | 0 | 4
  Indeterminate | 2 | 2 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -1.6, 95% CI 2-sided [-14.3 to 11.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -3.7, 95% CI 2-sided [-16.8 to 9.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 0.0, 95% CI 2-sided [-12.3 to 12.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -3.2, 95% CI 2-sided [-44.1 to 14.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the EOT Visit (Microbiological [Micro]-ITT Population)
Description: Clinical response was determined by the investigator at the EOT visit by assessing whether or not the participant met the clinical outcome of Clinical Success, Clinical Failure, or Indeterminate. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the EOT visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection at the EOT visit such that use of additional systemic antimicrobial therapy for the current infection was required. The clinical outcome was deemed as Indeterminate when the EOT visit was not completed.
Time Frame: EOT visit (within 1 to 2 days following the last dose of study drug i.e. up to approximately 9 days)
Population: The micro-ITT population consisted of all randomized participants who had a study-qualifying pre-treatment Baseline urine culture. A study-qualifying pretreatment Baseline culture was defined as a culture from a clean-catch urine sample which grew at least 1 and no more than 2 bacterial isolates at ≥ 10^5 colony forming unit (CFU)/mL each.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 25 | 34 | 23 | 5 | 30
Participants
  Clinical Success | 22 | 29 | 22 | 5 | 27
  Clinical Failure | 1 | 4 | 1 | 0 | 3
  Indeterminate | 2 | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -2.0, 95% CI 2-sided [-22.5 to 16.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -4.7, 95% CI 2-sided [-23.3 to 14.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 5.7, 95% CI 2-sided [-13.0 to 22.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 10.0, 95% CI 2-sided [-40.4 to 28.9] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the EOT Visit (CE-EOT Population)
Description: Clinical response was determined by the investigator at the EOT visit by assessing whether or not the participant met the clinical outcome of Clinical Success or Clinical Failure. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the EOT visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection at the EOT visit such that use of additional systemic antimicrobial therapy for the current infection was required. For the CE population, the clinical outcome was not deemed as indeterminate response.
Time Frame: EOT visit (within 1 to 2 days following the last dose of study drug i.e. up to approximately 9 days)
Population: The clinically evaluable (CE)-EOT population consisted of all ITT participants who completed the EOT visit, received test article, had a qualifying infection, an assessment of outcome, and met all other evaluability criterias.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 50 | 47 | 47 | 7 | 52
Participants
  Clinical Success | 47 | 42 | 47 | 7 | 48
  Clinical Failure | 3 | 5 | 0 | 0 | 4
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 1.7, 95% CI 2-sided [-10.0 to 13.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -2.9, 95% CI 2-sided [-16.2 to 9.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment Difference = 7.7, 95% CI 2-sided [-0.3 to 18.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatm,ent difference = 7.7, 95% CI 2-sided [-34.9 to 20.6] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the PTE Visit (CE-PTE Population)
Description: Clinical response was determined by the investigator at the PTE visit by assessing whether or not the participant met the clinical outcome of Clinical Success or Clinical Failure. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the PTE visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection or reappearance of signs and symptoms at or before the PTE visit such that use of additional systemic antimicrobial therapy for the current infection was required. For the CE population, the clinical outcome was not deemed as indeterminate response.
Time Frame: Day 14 (A PTE occurred on Day 14 ± 2 days after the participant's first dose of study drug)
Population: The clinically evaluable (CE)-PTE population consisted of all ITT participants who completed the PTE visit, received test article, had a qualifying infection, an assessment of outcome, and met all other evaluability criterias.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 49 | 46 | 47 | 7 | 49
Participants
  Clinical success | 45 | 41 | 46 | 7 | 45
  Clinical failure | 4 | 5 | 1 | 0 | 4
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 0.0, 95% CI 2-sided [-12.6 to 12.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -2.7, 95% CI 2-sided [-16.3 to 10.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 6.0, 95% CI 2-sided [-4.5 to 17.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 8.2, 95% CI 2-sided [-35.3 to 20.7] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the PTE Visit (Micro-ITT Population)
Description: Clinical response was determined by the investigator at the PTE visit by assessing whether or not the participant met the clinical outcome of Clinical Success, Clinical Failure or indeterminate. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the PTE visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection or reappearance of signs and symptoms at or before the PTE visit such that use of additional systemic antimicrobial therapy for the current infection was required. The clinical outcome was deemed as Indeterminate when the PTE visit was not completed.
Time Frame: Day 14 (A PTE occurred on Day 14 ± 2 days after the participant's first dose of study drug)
Population: The micro-ITT population consisted of consisted of all randomized participants who had a study-qualifying pre-treatment baseline urine culture. A study-qualifying pretreatment Baseline culture was defined as a culture from a clean-catch urine sample which grew at least 1 and no more than 2 bacterial isolates at ≥ 10^5 CFU/mL each.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 25 | 34 | 23 | 5 | 30
Participants
  Clinical success | 21 | 27 | 21 | 5 | 27
  Clinical failure | 2 | 5 | 2 | 0 | 3
  Indeterminate | 2 | 2 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -6.0, 95% CI 2-sided [-27.3 to 13.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -10.6, 95% CI 2-sided [-29.2 to 8.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment Difference = 1.3, 95% CI 2-sided [-19.0 to 19.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 10.0, 95% CI 2-sided [-40.4 to 28.9] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the Final Follow-up (FFU) Visit (ITT Population)
Description: Clinical response was determined by the investigator at the FFU visit by assessing whether or not the participant met the clinical outcome of Clinical Success, Clinical Failure, or Indeterminate. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the FFU visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection at the FFU visit such that use of additional systemic antimicrobial therapy for the current infection was required. The clinical outcome was deemed as Indeterminate when the FFU visit was not completed
Time Frame: FFU visit (A FFU occurred 30 to 37 days following the first dose of study drug)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 55 | 54 | 54 | 8 | 54
Participants
  Clinical success | 47 | 41 | 44 | 7 | 49
  Clinical failure | 6 | 7 | 7 | 0 | 5
  Indeterminate | 2 | 6 | 3 | 1 | 0
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -5.3, 95% CI 2-sided [-18.6 to 7.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -14.8, 95% CI 2-sided [-29.6 to -0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -9.3, 95% CI 2-sided [-23.2 to 4.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -3.2, 95% CI 2-sided [-44.1 to 14.7] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the FFU Visit (CE-FFU Population)
Description: Clinical response was determined by the investigator at the FFU visit by assessing whether or not the participant met the clinical outcome of Clinical Success or Clinical Failure. Clinical Success was defined as sufficient resolution of cystitis signs and symptoms at the FFU visit such that no additional systemic antimicrobial therapy was required for the current infection. Clinical Failure was defined as no apparent response to therapy or persistence of signs and symptoms of infection at the FFU visit such that use of additional systemic antimicrobial therapy for the current infection was required. For the CE population, the clinical outcome was not deemed as indeterminate response.
Time Frame: FFU visit (A FFU occurred 30 to 37 days following the first dose of study drug)
Population: The clinically evaluable (CE)-FFU Population consisted of all ITT participants who completed the FFU visit, received test article, had a qualifying infection, an assessment of outcome, and met all other evaluability criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 47 | 43 | 43 | 7 | 49
Participants
  Clinical success | 43 | 37 | 39 | 7 | 45
  Clinical failure | 4 | 6 | 4 | 0 | 4
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -0.3, 95% CI 2-sided [-13.1 to 12.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -5.8, 95% CI 2-sided [-20.7 to 7.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -1.1, 95% CI 2-sided [-15.1 to 11.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 8.2, 95% CI 2-sided [-35.3 to 20.7] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Number of Participants With an Investigator Assessment of Clinical Response at the FFU Visit (Micro-ITT Population)
Description: as for outcome 7
Time Frame: FFU visit (A FFU occurred 30 to 37 days following the first dose of study drug)
Population: The micro-ITT population consisted of all randomized participants who had a study-qualifying pre-treatment baseline urine culture. A study-qualifying pretreatment Baseline culture was defined as a culture from a clean-catch urine sample which grew at least 1 and no more than 2 bacterial isolates at ≥ 10^5 CFU/mL each.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 25 | 34 | 23 | 5 | 30
Participants
  Clinical success | 21 | 26 | 20 | 5 | 27
  Clinical failure | 2 | 6 | 3 | 0 | 3
  Indeterminate | 2 | 2 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -6.0, 95% CI 2-sided [-27.3 to 13.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -13.5, 95% CI 2-sided [-32.4 to 5.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -3.0, 95% CI 2-sided [-25.7 to 15.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 10.0, 95% CI 2-sided [-40.4 to 28.9] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Participants With a Microbiological Response at the EOT Visit (Micro-ITT Population)
Description: Microbiological response was determined programmatically at the EOT visit by assessing whether or not the participant met the microbiological outcome of Favorable, Unfavorable, or Indeterminate. Favorable microbiological outcomes included eradication and presumed eradication i.e., urine specimen showed absence of the original baseline pathogen or the baseline pathogen grew at <10^4 CFU/mL at visit. Unfavorable microbiological outcome included persistence i.e. urine culture showed continued presence (defined as ≥10^4 CFU/mL) of the original baseline pathogen(s) at visit. The microbiological outcome was deemed as Indeterminate when the urine specimen was not available to culture or the culture result was not interpretable.
Time Frame: EOT visit (within 1 to 2 days following the last dose of study drug i.e. up to approximately 9 days)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 25 | 34 | 23 | 5 | 30
Participants
  Favorable | 18 | 27 | 17 | 5 | 28
  Unfavorable | 5 | 6 | 6 | 0 | 1
  Indeterminate | 2 | 1 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -21.3, 95% CI 2-sided [-44.1 to -1.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -13.9, 95% CI 2-sided [-32.2 to 4.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -19.4, 95% CI 2-sided [-43.1 to 1.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 6.7, 95% CI 2-sided [-43.8 to 23.2] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Participants With a Microbiological Response at the EOT Visit (ME-EOT Population)
Description: Microbiological response was determined programmatically at the EOT visit by assessing whether or not the participant met the microbiological outcome of Favorable or Unfavorable. Favorable microbiological outcomes included eradication and presumed eradication i.e., urine specimen showed absence of the original baseline pathogen or the baseline pathogen grew at <10^4 CFU/mL at visit. Unfavorable microbiological outcome included persistence i.e. urine culture showed continued presence (defined as ≥10^4 CFU/mL) of the original baseline pathogen(s) at visit. For the ME population, the microbiological outcome was not deemed as indeterminate response.
Time Frame: EOT visit (within 1 to 2 days following the last dose of study drug i.e. up to approximately 9 days)
Population: The microbiologically evaluable (ME)-EOT population consisted of participants in the micro-ITT and CE-EOT populations who had a study-qualifying pre-treatment baseline urine culture with 1 or 2 uropathogens at ≥ 10^5 CFU/mL.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 22 | 31 | 22 | 5 | 29
Participants
  Favorable | 18 | 25 | 16 | 5 | 28
  Unfavorable | 4 | 6 | 6 | 0 | 1
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -14.7, 95% CI 2-sided [-37.2 to 3.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -15.9, 95% CI 2-sided [-34.3 to 1.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -23.8, 95% CI 2-sided [-46.9 to -4.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 3.4, 95% CI 2-sided [-48.5 to 19.7] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Number of Participants With a Microbiological Response at the PTE Visit (Micro-ITT Population)
Description: Microbiological response was determined programmatically at the PTE visit by assessing whether or not the participant met the microbiological outcome of Favorable, Unfavorable, or Indeterminate. Favorable microbiological outcomes included eradication and presumed eradication i.e., urine specimen showed absence of the original baseline pathogen or the baseline pathogen grew at <10^4 CFU/mL at visit. Unfavorable microbiological outcome included persistence i.e. urine culture showed continued presence (defined as ≥10^4 CFU/mL) of the original baseline pathogen(s) at visit. The microbiological outcome was deemed as Indeterminate when the urine specimen was not available to culture or the culture result was not interpretable.
Time Frame: Day 14 (A PTE occurred on Day 14 ± 2 days after the participant's first dose of study drug)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 25 | 34 | 23 | 5 | 30
Participants
  Favorable | 14 | 20 | 15 | 4 | 23
  Unfavorable | 8 | 11 | 8 | 1 | 6
  Indeterminate | 3 | 3 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -20.7, 95% CI 2-sided [-45.1 to 6.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -17.8, 95% CI 2-sided [-40.2 to 5.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -11.4, 95% CI 2-sided [-36.8 to 14.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 3.3, 95% CI 2-sided [-47.0 to 33.2] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Number of Participants With a Microbiological Response at the PTE Visit (ME-PTE Population)
Description: Microbiological response was determined programmatically at the PTE visit by assessing whether or not the participant met the microbiological outcome of Favorable or Unfavorable. Favorable microbiological outcomes included eradication and presumed eradication i.e., urine specimen showed absence of the original baseline pathogen or the baseline pathogen grew at <10^4 CFU/mL at visit. Unfavorable microbiological outcome included persistence i.e. urine culture showed continued presence (defined as ≥10^4 CFU/mL) of the original baseline pathogen(s) at visit. For the ME population, the microbiological outcome was not deemed as indeterminate response.
Time Frame: Day 14 (A PTE occurred on Day 14 ± 2 days after the participant's first dose of study drug)
Population: The ME-PTE population consisted of participants in the micro-ITT and CE-PTE populations who had a study-qualifying pre-treatment baseline urine culture with 1 or 2 uropathogens at ≥ 10^5 CFU/mL.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 20 | 29 | 21 | 5 | 28
Participants
  Favorable | 13 | 20 | 14 | 4 | 22
  Unfavorable | 7 | 9 | 7 | 1 | 6
Statistical Analysis 1: Comparison: Omadacycline 300/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -13.6, 95% CI 2-sided [-40.4 to 13.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Omadacycline 450/300 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -9.6, 95% CI 2-sided [-32.7 to 14.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Omadacycline 450/450 Once Every 24 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = -11.9, 95% CI 2-sided [-38.2 to 14.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Omadacycline 450/450 Once Every 12 Hours vs Nitrofurantoin 100/100 Once Every 12 Hours; Test type: Non-Inferiority — Non-inferiority margin for comparison of the doses was set at 10%; Treatment difference = 1.4, 95% CI 2-sided [-50.3 to 30.9] — [estimate comment as in outcome 1, analysis 1]

14. Other Pre Specified Outcome: Number of Participants With Resolution of All Urinary Tract Infection (UTI) Signs and Clinical Symptoms at PTE Visit (ITT Population)
Description: Participants recorded their assessments using the UTI Symptoms Assessment (UTISA) questionnaire, a 14-item questionnaire that assessed the levels of 'severity' and 'bothersomeness' for seven UTI signs and symptoms: Frequency, Urgency, Pain/burning on urination, Incomplete voiding, Pain in pelvic area, Low back pain, and Blood in urine. The sub-scale responses were recorded as 'did not have', 'mild', 'moderate', and 'severe' for 'severity'; and 'not at all', 'a little', 'moderately', and 'a lot' for 'bothersomeness', both scored 0-3. Total scores were calculated by summing the non-missing scores of the 7 items, divided by the number of non-missing items, and then multiplied by 7. For each sub-scale, the total score ranged from 0 (least Severe/ least bothersome) and 21 (worst severity/most bothersome). Number of participants with resolution of all symptoms, without occurrence of new symptoms is reported. Resolution was defined as absence of all baseline symptoms.
Time Frame: Day 14 (A PTE occurred on Day 14 ± 2 days after the participant's first dose of study drug)
Population: The ITT population consisted of all randomized participants regardless of whether or not the participant received study drug. Participants who completed the PTE visit were analyzed for this end point.
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 51 | 47 | 49 | 7 | 51
Participants | 33 | 30 | 32 | 6 | 34

15. Other Pre Specified Outcome: Number of Participants With No Worsening and Absence of New UTI Signs and Clinical Symptoms at PTE Visit (ITT Population)
Description: Participants recorded their assessments using the UTI Symptoms Assessment (UTISA) questionnaire, a 14-item questionnaire that assessed the levels of 'severity' and 'bothersomeness' for seven UTI signs and symptoms: Frequency, Urgency, Pain/burning on urination, Incomplete voiding, Pain in pelvic area, Low back pain, and Blood in urine. The sub-scale responses were recorded as 'did not have', 'mild', 'moderate', and 'severe' for 'severity'; and 'not at all', 'a little', 'moderately', and 'a lot' for 'bothersomeness', both scored 0-3. Total scores were calculated by summing the non-missing scores of the 7 items, divided by the number of non-missing items, and then multiplied by 7. For each sub-scale, the total score ranged from 0 (least Severe/ least bothersome) and 21 (worst severity/most bothersome). Number of participants with no worsening and absence of new UTI signs and clinical symptoms is reported. No worsening meant that each question score is same or better at post baseline.
Time Frame: Day 14 (A PTE occurred on Day 14 ± 2 days after the participant's first dose of study drug)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
Number analyzed (Participants) | 51 | 47 | 49 | 7 | 51
Participants | 50 | 45 | 45 | 7 | 50

ADVERSE EVENTS:
Time Frame: Up to approximately 37 days
Description: A treatment-emergent adverse event was defined as any adverse event that newly appeared, increased in frequency, or worsened in severity on or after the initiation of the study drug.
Arm/Group | Omadacycline 300/300 Once Every 24 Hours | Omadacycline 450/300 Once Every 24 Hours | Omadacycline 450/450 Once Every 24 Hours | Omadacycline 450/450 Once Every 12 Hours | Nitrofurantoin 100/100 Once Every 12 Hours
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54 | 0/54 | 0/8 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 1/54 | 0/8 | 0/54
Other Adverse Events (participants affected / at risk) | 16/55 | 13/54 | 15/54 | 4/8 | 9/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline 300/300 Once Every 24 Hours (N=55) | Omadacycline 450/300 Once Every 24 Hours (N=54) | Omadacycline 450/450 Once Every 24 Hours (N=54) | Omadacycline 450/450 Once Every 12 Hours (N=8) | Nitrofurantoin 100/100 Once Every 12 Hours (N=54)
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline 300/300 Once Every 24 Hours (N=55) | Omadacycline 450/300 Once Every 24 Hours (N=54) | Omadacycline 450/450 Once Every 24 Hours (N=54) | Omadacycline 450/450 Once Every 12 Hours (N=8) | Nitrofurantoin 100/100 Once Every 12 Hours (N=54)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 2
Nausea (Gastrointestinal disorders) | 12 | 8 | 10 | 4 | 5
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 4 | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
An additional treatment group (omadacycline 450/450 once every 12 hours) was added with Protocol Amendment 2. However, the majority of enrollment was completed by this time, and therefore, fewer participants were enrolled in this group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication and require the removal of confidential information.

DOCUMENTS (2):
  • Study Protocol (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT03425396/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03425396/SAP_001.pdf